CLINICAL TRIAL: NCT05856214
Title: Effect of Couple-Based Violence Prevention Education on Intimate Partner Violence in Hadiya Zone, Southwest Ethiopia
Brief Title: Effect of Couple Based Violence Prevention Education on Intimate Partner Violence During Pregnancy in Southern, Ethiopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: Wachemo University (Other)
Responsible Party: Principal Investigator, Zeleke Dutamo, Primary Investigator, Jimma University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Couple-Based Education
Record Dates: First submitted 2023-03-30; First posted 2023-05-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Intimate Partner Violence
Keywords: Intimate partner violence; Hadiya zone; Southwest Ethiopia

STUDY DESIGN:
Intervention Model Description: Single group assignment: intervention group vs Control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Couple-based violence prevention education(CBVPE) (Experimental): Couples in the intervention group will receive trainings on gender based violence, intimate partner violence, Consequences of violence during pregnancy, common triggers of intimate partner violence, a healthy relationship in marriage ,couples communication and conflict management
  Interventions: Behavioral: Couple-Based Violence Prevention education(CBVPE)

INTERVENTIONS:
Behavioral: Couple-Based Violence Prevention education(CBVPE) — Couples in the intervention group will receive training on violence against women including intimate partner violence, types, and consequences of intimate partner violence during pregnancy, managing triggers of intimate partner violence, healthy relationships, the role of male partners during pregnancy, and couples communication and problem-solving skills. Training will be provided every fourth week by trained health extension workers for consecutive six months.

SUMMARY:
A significant proportion of women in Ethiopia suffer from violence by their intimate partner during pregnancy(IPVp), which has adverse maternal and newborn outcomes. Intervention addressing their intimate partners are not well-studied, particularly in Ethiopian setting. The investigators use a cluster randomized control study to evaluate the effectiveness of Couple-Based Violence Prevention Education(CBVPE). CBVPE is an intervention aimed to improve experience of violence during pregnancy, male partners knowledge, attitudes and controlling behavior towards intimate partner violacein this study kebeles found under each districts will be used as clusters. Sixteen clusters will be randomly assigned into one of two arms, each comprised of 216 couples. A total of 864 participants (432 pregnant women and 432 their male partners will be recruited for the study. women in the control group will receive the usual care provided by Health Extension Workers(HEWs), which is routine care. The intervention arm, wife and husband will be exposed to CBVPE that explores maternal health, intimate partner violence, adverse effects of violence during pregnancy, triggers of IPV, managing triggers of IPV, problem solving skills and health relationship. Our hypothesis is that CBVPE is superior to routine care in reducing and /or controlling intimate partner violence during pregnancy in HadiyaZone, Southwest Ethiopia. Structured interviewer administered questionnaire will be used to collect data at base-line and end-line.

DETAILED DESCRIPTION:
Violence during pregnancy is a possible risk to not only the pregnant mother but also the risk to that unborn child. IPV during pregnancy is associated with adverse maternal outcomes including emotional distress, depression, anxiety, insufficient or inconsistent prenatal care, inadequate gestational weight gain, higher rates of smoking, alcohol use, and mortality. In Ethiopia, intimate partner violence is one of the hidden epidemics, that needs appropriate intervention strategy. Couples in intervention arm 1 will be exposed to CBVPE, which explores intimate partner violence, consequences of violence during pregnancy, common triggers of IPV during pregnancy, the role of male partners in pregnancy, healthy relationships, and problem-solving skills. Couples in control arm 2, will receive the usual care provided by the Health Extension Workers. Our hypothesis is that women in intervention arm 1 will report less experience of intimate partner violence than participants in arm 2, the control group. Data will be collected at baseline and end line using a structured questionnaire. The study has the following specific objectives

1. To evaluate the effect of couple-based violence prevention education on male partners' knowledge, attitudes, and controlling behavior towards IPV during pregnancy
2. To compare the effect of couple-based violence prevention education on the experience of IPV during pregnancy
3. To Compare the effect of couple-based violence prevention education on women's autonomy and self-efficacy

ELIGIBILITY:
Inclusion Criteria:

* Coupe whose wife is pregnant (trimester)
* Couple whose wife has at least one live birth
* Couple who lived in the study area at least six months before the study
* Couple whose wife's inter-pregnancy interval is less than two years
* Couple willing to be visited at home

Exclusion Criteria:

* Couple having a severe medical illness
* Couple with hearing or communication problems
* Couple with a plan to move out from the intervention and control clusters in the next 8 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 852 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of women who experience intimate partner violence during pregnancy | 8 months
  WHO Multi-country Study on Women's Health and Domestic Violence against Women questionnaire is adapted to assess intimate partner violence (IPV).
  Physical violence: the intentional use of physical forces by the husband (Slap, push, shove or pull hair, kick, drag or beat, attempt to choke or burn on purpose, threaten to use or actually use a gun, knife, or another weapon) Sexual violence: when a husband forces his wife to have sexual intercourse with him when she doesn't want to, forces her with threats, in any other way to perform sexual acts she does not want, and/or physically forces her to perform any other sexual acts she does not want to Psychological violence: when the husband says or does something to humiliate his wife in front of another person and /or threatens to hurt or harm someone she cares about and/or insult or make her feel bad about herself. IPV is when the woman experiences any physical and/or sexual and/or psychological violence in combination during pregnancy

SECONDARY OUTCOMES:
The difference in the proportion of couples' attitudes, and husband's controlling behavior(AC) toward intimate partner violence | 8 months
  WHO Multi-country Study on Women's Health and Domestic Violence against Women questionnaire is adapted to assess couples' attitudes towards IPV during pregnancy. Couples will be asked whether a husband is justified in hitting or beating his wife in 5 scenarios: If the wife goes out without telling the husband, if the wife neglects the children, if the wife argues with the husband if the wife refuses to have sex with husband, and if she burns the food. The response will be coded as '1' if the participant agrees with at least one attitude question, otherwise will be coded as '0' Couples will be asked six controlling questions. If the husband: is jealous if she talks with other men, accuses her of unfaithfulness, does not permit her to meet her friends, tries to limit her contact with family, insists on knowing where she is, and does not trust her with money. Couples who responded "yes" to one or more of the control questions will be coded as 1. Otherwise, it will be coded 'no' as 0.

CONTACTS AND LOCATIONS:
Overall Officials: Zeleke D Agde, MPH, Principal Investigator — Department of population and family studies, Institute of Health, Jimma University, Ethiopia; Muluemebet A Wordofa, professor, Study Chair — Department of population and family studies, Institute of health, Jimma University, Ethiopia; Nega A Kassa, Professor, Study Director — College of Medical and Health Sciences, Haramaya University, Ethiopia; Jeanette H Magnus, Professor, Study Director — University of Oslo
Locations (1):
- 1st Benara Health post, Hosa’ina, Central Ethiopia/Hadiya Zone, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data(IPD) will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting August,2024

REFERENCES:
- [Derived] Agde ZD, Magnus JH, Assefa N, Wordofa MA. Effects of couple-based violence prevention education on male partners' knowledge, attitudes and controlling behavior related to intimate partner violence in rural Ethiopia: a cluster randomized controlled trial. Front Public Health. 2025 Mar 10;13:1506459. doi: 10.3389/fpubh.2025.1506459. eCollection 2025. PMID 40129596
- [Derived] Agde ZD, Magnus JH, Assefa N, Wordofa MA. Effectiveness of couple-based violence prevention education in reducing intimate partner violence during pregnancy in rural Ethiopia: A cluster randomized controlled trial. PLoS One. 2025 Jan 17;20(1):e0317667. doi: 10.1371/journal.pone.0317667. eCollection 2025. PMID 39823488
- [Derived] Agde ZD, H Magnus J, Assefa N, Wordofa MA. The protocol for a cluster randomized controlled trial to evaluate couple-based violence prevention education and its ability to reduce intimate partner violence during pregnancy in Southwest Ethiopia. PLoS One. 2024 May 13;19(5):e0303009. doi: 10.1371/journal.pone.0303009. eCollection 2024. PMID 38739581